CLINICAL TRIAL: NCT06448663
Title: Targeting the Gut to Improve Seizure Control in CDD
Brief Title: Targeting the Gut to Improve Seizure Control in CDKL5 Deficiency Disorder (CDD)
Acronym: NUTRIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Telethon (Other); Kolfarma s.r.l. - Italy (Unknown)
Responsible Party: Principal Investigator, Aglaia Vignoli, Professor, University of Milan
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GSA23G001
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: CDKL5
Keywords: epilepsy, gut microbiota, sleep disorders
MeSH Terms: conditions — Epilepsy; Sleep Wake Disorders | interventions — Lactalbumin; fructooligosaccharide; Inulin; Butyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDD arm (Experimental): This is a 32-week pilot, single site, cross-over trial of alpha-lactalbumin+ inulin + fructo-oligosaccharides vs alpha-lactalbumin + sodium butyrate + inulin + fructo-oligosaccharides. Periods I and II of the study are 12-week long together with a 4-week washout period.
  Interventions: Dietary Supplement: alpha-lactalbumin, fructooligosaccharides, inulin; Dietary Supplement: alpha-lactalbumin, sodium butyrate, fructooligosaccharides, inulin

INTERVENTIONS:
Dietary Supplement: alpha-lactalbumin, fructooligosaccharides, inulin — The first round supplementation will be administered for 3-month period (i.e. 12 weeks). One dose/day (2g sachet) is intended to be administered orally once a day after dissolving in water.
  At the scheduled visits/phone contacts [i.e., baseline, 12 weeks, and 16 weeks (post washout)], seizure frequency and entity of the critical episodes will be recorded. Gut microbiome characterization, clinical scales and dietary intake will be assessed.
Dietary Supplement: alpha-lactalbumin, sodium butyrate, fructooligosaccharides, inulin — The second round supplementation will be administered for 3-month period (i.e. 12 weeks). For participants weighing <30 kg, a 4 g dose (i.e., one 4 g sachet) is intended to be administered orally once a day after dissolving in water. For participants weighing ≥30 kg, a 4 g dose (i.e., 4 g sachets) is intended to be administered orally twice a day (12h interval) after dissolving in water.
  At the scheduled visits/phone contacts [i.e., 28 weeks and 32 weeks (post washout)], seizure frequency and entity of the critical episodes will be recorded. Gut microbiome characterization, clinical scales and dietary intake will be assessed.

SUMMARY:
Standard anti-seizure medications have limited efficacy in seizure control in cyclin-dependent kinase-like 5 deficiency disorder (CDD).

The study will investigate whether targeting the gut-microbiota-brain axis in CDD patients can alleviate seizures and ameliorate other comorbidities.

DETAILED DESCRIPTION:
CDD is a neurodevelopmental condition characterized by infantile-onset epilepsy, developmental delays, intellectual and motor disabilities, sleep disturbances, and cortical visual impairment. Currently, there is no treatment for CDD, and epilepsy is a prominent and severe feature of the disorder. Standard anti-seizure medications have limited efficacy in seizure control, leading to detrimental effects on cognitive and motor development in CDD.

The gut-brain axis has gained attention in epilepsy research, prompted by evidence of gastrointestinal (GI) symptoms in people with epilepsy. Studies have demonstrated significant changes in gut microbial composition in animal models and between individuals with epilepsy and healthy subjects. Notably, CDD patients experience GI problems, and we discovered that they exhibit alterations in their gut microbiota compared to healthy individuals. The study will investigate whether supplementing CDD patients with alpha-lactalbum and prebiotics alone or with post-biotics can improve neurological features and modulate microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of CDD and demonstrated CDKL5 pathogenic variant; drug-resistant seizures; ensured participation of a caregiver; willingness to sign the informed consent.

Exclusion Criteria:

organic GI disorders (i.e., food allergies, celiac disease); special diets; percutaneous endoscopic gastrostomy tube; use of antibiotics or probiotics in the previous month.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Epilepsy | Change at 3 months from baseline of each round of supplementation
  to evaluate the number of CDD patients considered treatment responders (seizure reduction ≥50%, ≥75% or ≥100% from baseline in monthly seizure counts) during the 12- week treatment period in 1st and 2nd round of supplementation

SECONDARY OUTCOMES:
Gut microbiota | Change at 3 months from baseline of each round of supplementation
  to evaluate indicator species that could help as biomarkers for guiding clinicians to choose the intervention with the most likelihood of improve patient quality of life.
Sleep disturbances | Change at 3 months from baseline of each round of supplementation
  Decreased Sleep SDSC scale (max score=125) by at least 5%
gastrointestinal discomfort | Change at 3 months from baseline of each round of supplementation
  Decrease GISI scale (max score = 17), by at least 2 points

OTHER OUTCOMES:
Clinical features | Change at 3 months from baseline of each round of supplementation
  Clinical Global Impression of Change (CGIC), ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change] decrease of at least 1 point
Parental stress | Change at 3 months from baseline of each round of supplementation
  Caregiver burden by Parenting Stress Index (PSI-SF); clinically significance > 85%, decrease by at least 5%

CONTACTS AND LOCATIONS:
Overall Officials: Aglaia Vignoli, MD, Principal Investigator — University of Milan
Locations (1):
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borghi E, Xynomilakis O, Ottaviano E, Ceccarani C, Vigano I, Tognini P, Vignoli A. Gut microbiota profile in CDKL5 deficiency disorder patients. Sci Rep. 2024 Mar 28;14(1):7376. doi: 10.1038/s41598-024-56989-0. PMID 38548767
- [Derived] Triva F, Borghi E, Marsiglia MD, Ottaviano E, Ricci E, Tognini P, Montecucco M, Vignoli A. Targeting the gut to improve seizure control in CDKL5 deficiency disorder (CDD): study protocol for a single-arm, open-label clinical trial. Front Neurol. 2025 Oct 28;16:1642329. doi: 10.3389/fneur.2025.1642329. eCollection 2025. PMID 41230376